CLINICAL TRIAL: NCT01996280
Title: A Randomized Clinical Trial of Culturally Tailored Motivational Interviewing
Brief Title: A Randomized Clinical Trial of Culturally Tailored MI
Acronym: CTMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PA-10-100
Record Dates: First submitted 2013-06-17; First posted 2013-11-27 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Placebo Comparator): The MI is a single brief motivational intervention lasting 1.5 hours that includes MI structured strategies tailored to the patient's readiness to change such as: the Typical Day exercise, the use of personal feedback reports (e.g., normative feedback about their drinking), discussions about the pros and cons of use, and completion of a change plan. The MI is designed to follow MI principles of invoking autonomy and emphasizing collaboration with the interventionist.
  Interventions: Behavioral: Motivational Interviewing
- Culturally Tailored MI (Experimental): The CTMI is a single brief motivational interview lasting 1.5 hours. It follows the same sequence of structured strategies as the MI, but the focus of the components is different. CTMI has augmented some of the components with culturally relevant material, including discussion about acculturation stress. The CTMI components are culturally tailored to address relevant concerns and issues. There are also culturally tailored feedback elements in the CTMI, such as ethnic normative feedback about drinking. To control for time across conditions, interventionists are instructed to select CTMI components based on participant interests, not the entire array of components.
  Interventions: Behavioral: Culturally Tailored MI

INTERVENTIONS:
Behavioral: Motivational Interviewing — The MI is a single brief motivational intervention lasting 1.5 hrs. The MI includes MI structured strategies tailored to the patient's readiness to change such as: the Typical Day exercise, the use of personal feedback reports (e.g., normative feedback about their drinking), discussions about the pros and cons of use, and completion of a change plan; It is designed to follow MI principles of invoking autonomy and emphasizing collaboration with the interventionist.
  Arms: Motivational Interviewing
Behavioral: Culturally Tailored MI — CTMI is a single brief motivational intervention lasting 1.5hrs. The CTMI follows the same sequence of structured strategies as the MI arm, and while the components in CTMI and MI are parallel, the focus within them is different. CTMI components culturally relevant material, such as acculturation stress. The CTMI components, which are MI structured strategies, are culturally tailored to address relevant concerns and issues. There are also culturally tailored feedback element, such as ethnic normative feedback related to drinking.
  Arms: Culturally Tailored MI

SUMMARY:
Culturally-tailored empirically-based interventions are needed because Latinos suffer a greater burden of alcohol-related health disparities and negative social consequences compared to other racial/ethnic groups, are less likely to initiate and to remain in treatment, and are more likely to live in communities with a high density of alcohol outlets. Pilot data from the PI's (New Investigator) K award (AA014905), which will serve as the basis for the current proposed larger-scale study, demonstrated that culturally tailored motivational interviewing (CTMI) outperformed motivational interviewing (MI) that was not tailored to the needs of Latino heavy drinkers. The public health impact of this study will be to develop a program of early screening and brief intervention to reduce hazardous drinking among Latinos, to minimize the burden of illness and social consequences that disproportionately affect Latino communities.

DETAILED DESCRIPTION:
The proposed R01 research, in response to PA 10-100, "Alcohol Use Disorders: Treatment, Services Research, and Recovery", addresses the PA priority: Treatment for Health Disparities/Special Populations. Latinos, the largest and fastest growing ethnic group in the United States (U.S.), representing 14% of the population (1), are expected to grow to nearly 29% of the population by 2050 (2-3). Like many immigrant groups adapting to U.S. culture, Latinos adopt the health behaviors of the mainstream population, such as hazardous drinking (4-6). Hazardous drinking is a pattern of drinking associated with increased alcohol related problems: injuries, violence, sexually transmitted diseases (7-15), and increased risk for developing an alcohol use disorder (abuse or dependence) (7, 10, 16). Latinos report a disproportionately greater burden of illness, injuries, workplace and legal problems (17-21) as a result of their alcohol consumption than other racial ethnic groups, including an elevated risk for alcohol-involved motor vehicle crashes and fatalities (20, 22).

Early intervention prevents the need for more costly and complex alcohol treatment (23). According to the National Academy of Sciences, dissemination of empirically-based interventions that are culturally tailored is particularly needed among Latinos (23-24) because they suffer alcohol-related health disparities (18-20, 25-26) and because alcohol treatment utilization rates are lower among Latinos than among other minority racial/ethnic groups or Whites (27-29). Although evidence suggests that culturally tailored addiction treatment improves retention and treatment outcomes (30-31), progress in the field has been limited by the lack of prospective clinical trials comparing tailored to non-tailored treatment (23). The PI's (New Investigator) funded K award (AA014905) provided important pilot data demonstrating that culturally tailored motivational interviewing (CTMI) outperformed un-tailored motivational interviewing (MI). This study will be the basis for the current proposed study, which is a larger scale version of the pilot. The culturally tailored MI maintained MI components. The key modification in our Social Contextual Model of Cultural Tailoring was to tailor the MI to incorporate important acculturation stressors (32-33): limited financial resources and opportunities, loss of social networks, discrimination (34-38), and changing cultural values. The proposed study will investigate acculturation stress (39) as an influence on the relationship between acculturation and alcohol consumption behavior and treatment outcomes. Efforts will help build a comprehensive model of how acculturation stressors influence drinking behavior among Latinos (40). The CTMI is also a needed effort to tailor treatment to drinkers who experience the burden of multiple social contextual sources of disadvantage, including poverty, discrimination, and acculturation stress (40).

Because the original pilot study goal was to isolate and test the effects of tailoring treatment, it was delivered in English. The current proposal extends the tailored treatment to Spanish-speaking Latinos. Providing the tailored treatment in Spanish addresses a major clinical need and increases external generalizability. The study's public health impact will be to provide early screening and brief intervention to reduce hazardous drinking among Latinos in communities that lack such services. By providing early screening and intervention, we hope to minimize the burden of illness and social consequences that disproportionately affect Latino communities. Impact on field: will be to contribute to an understanding of whether culturally tailored motivational intervention enhances treatment efficacy for Latinos compared to un-tailored treatment. Another contribution will be to explore the effects of translating and of tailoring MI. Short term goals are to compare the efficacy of an evidenced-based treatment, MI, against a culturally adapted version of MI among Latinos. Long term goals are to disseminate an easily trainable, conceptual model of culturally tailored empirically-based substance abuse treatment, understand how acculturation processes confer risk for increased hazardous drinking among Latinos, and to inform further tailoring of treatments for multiple stressors, including acculturation stress.

Research Hypotheses:

Primary Aim 1: Treatment Main Effect. Determine the efficacy of standard motivational interviewing (MI) compared to culturally tailored MI (CTMI) at two, six, and twelve month follow-up. We hypothesize that CTMI participants will report fewer alcohol-related negative consequences and fewer heavy drinking days at follow-up vs. MI participants.

Primary Aim 2: Explore acculturation stress as a moderator of alcohol treatment outcomes for Latinos. We hypothesize that among participants with high acculturation stress, those in CTMI will improve more over time than those in MI (at 6 months). We also hypothesize that among those who receive CTMI, those with high acculturation stress may show greater improvement over time (at six months) than those with low acculturation stress.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for hazardous drinking (greater than or equal to 5/4 per occasion for males/females), two or more times in the past 30 days.
* Latino
* Are not currently in any substance use treatment program for alcohol use disorder, nor have been in the past year.
* 18-65 years old
* Able to speak English or Spanish

Exclusion Criteria:

* Psychotic symptoms, as evidenced by hallucinations or delusions.
* Cognitive impairment, as evidenced by inability to understand informed consent. a. To determine comprehension, a research assistant will read informed consent aloud and will ask 3 questions

  1. Is the study voluntary
  2. Can he/she drop out at any time
  3. Will there be study follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2014-08-26 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Frequency of Heavy Drinking Days | Baseline, 3-, 6-, and 12-month follow-up
  The frequency of heavy drinking days will be assessed using a 90 day Timeline Follow Back (TLFB) collected at baseline prior to study intervention. TLFB will be administered again at the 3-, 6-, and 12-month follow up periods. Changes in frequency of heavy drinking days will be assessed across all study time points.

SECONDARY OUTCOMES:
Change in Frequency of Alcohol-Related Negative Consequences | Baseline, 3-, 6-. 12-month follow up
  Frequency of alcohol-related consequences will be assessed using the Drinker Inventory of Consequences (DrInC) and its' five subscales, as well as the Drinking and Driving Scale. The DrInC will be administered at baseline, 3-, 6-, and 12-month follow up whereas the Drinking and Driving scale will be administered at baseline and again at the 12-month follow up session. Changes in the frequency of reported negative alcohol-related consequences will be examined across these time points.

CONTACTS AND LOCATIONS:
Overall Officials: Christina S Lee, Ph.D, Principal Investigator — Northeastern University
Locations (2):
- United States (2):
  - Northeastern University, Boston, Massachusetts
  - South End Community Health Center, Boston, Massachusetts

REFERENCES:
- [Derived] Rosales R, Lee CS, Cortes D, Caetano R, Rohsenow DJ, Lopez SR, Colby SM. Development and Evaluation of a Measure of Drinking Behavior in Response to Acculturation Stressors for Latinx Adults Entering Alcohol Treatment. J Subst Use Addict Treat. 2023 Dec;155:208936. doi: 10.1016/j.josat.2022.208936. Epub 2023 Jan 13. PMID 38434594
- [Derived] Hai AH, Lee CS, Zhou C, Delva J. Culturally adapted motivational interviewing's effects on drinking in response to immigration and acculturation stressors among Latinx adults with heavy drinking problems. J Subst Use Addict Treat. 2023 Jul;150:209061. doi: 10.1016/j.josat.2023.209061. Epub 2023 May 6. PMID 37156426
- [Derived] Lee CS, Colby SM, Rohsenow DJ, Martin R, Rosales R, McCallum TT, Falcon L, Almeida J, Cortes DE. A randomized controlled trial of motivational interviewing tailored for heavy drinking latinxs. J Consult Clin Psychol. 2019 Sep;87(9):815-830. doi: 10.1037/ccp0000428. PMID 31403817
- [Derived] Lee CS, Almeida J, Colby SM, Tavares T, Rohsenow DJ. Acculturation, hazardous drinking and depressive symptomatology among Hispanics enrolled in a clinical trial. Addict Res Theory. 2016 Jan 1;24(1):69-79. doi: 10.3109/16066359.2015.1072517. Epub 2015 Jul 28. PMID 26819573